CLINICAL TRIAL: NCT04721119
Title: Comparison of the Effectiveness of Adductor Canal Block Versus Combination of Adductor Canal Block and Local Infiltration Analgesia: A Randomized Controlled Trial of the Effect on Postoperative Analgesia and Motor Power
Brief Title: Comparing Adductor Canal Block and Adductor Canal Block-Local Infiltration Analgesia for Post-operative Pain Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2382
Record Dates: First submitted 2020-08-19; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: ACL Tear; ACL; ACL Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local Infiltration Anesthetic (Experimental): This group of patients will receive the local infiltration anesthetic only.
  Interventions: Procedure: Local Infiltration Anesthetic
- Local Infiltration Anesthetic + Adductor Canal Block (Experimental): This group of patients will receive the local infiltration anesthetic and adductor canal block combination.
  Interventions: Procedure: Local Infiltration Anesthetic + Adductor Canal Block

INTERVENTIONS:
Procedure: Local Infiltration Anesthetic — For the local infiltration anesthetic, patients will receive 20 cc of 0.5% ropivacaine, by intra-articular injection performed by the surgeon. The injection is done at the end of the surgical procedure, after suturing the incision.
  Arms: Local Infiltration Anesthetic
Procedure: Local Infiltration Anesthetic + Adductor Canal Block — For the local infiltration anesthetic, patients will receive 20 cc of 0.25% ropivacaine, by intra-articular injection performed by the surgeon. The injection is done at the end of the surgical procedure, after suturing the incision. For the adductor canal block, patients will receive 20 cc of 0.25% ropivicaine, through injection performed by the anesthesiologist. The injection is done under the sartorius muscle, in mid-thigh, using ultrasound guidance.
  Arms: Local Infiltration Anesthetic + Adductor Canal Block

SUMMARY:
Anterior cruciate ligament (ACL) reconstruction is one of the most commonly performed surgeries amongst young orthopedic surgery patients. Optimal post-operative pain control helps to reduce the opioid burden and to improve the patient's experience. Regional anesthesia, such as the femoral nerve block (FNB) and adductor canal block (ACB), are commonly used for post-operative pain control after surgery. The ACB has replaced the FNB. This is because the ACB targets the femoral nerve, while avoiding the numbing effects on quadricep muscle strength that make it difficult to move the leg. Another form of pain control is local infiltration anesthesia (LIA), which directly blocks pain in the knee. Similar to the ACB, it avoids the numbing effects on the quadricep muscle.This can help improve patient safety and experience by reducing risks of falls and allowing the patient to move earlier. This can also be associated with decreased time in the hospital and decreased costs. Technically, it is less complex and can be done the shorter period of time.

The purpose of this study is to refine the pain management technique following anterior cruciate ligament surgery. More specifically, the aim of this study is to evaluate the effects of LIA alone, and a LIA-ACB combination on post-operative pain and thigh muscle strength.

ELIGIBILITY:
Inclusion Criteria:

* English speaking or any other language with possibility of adequate translation
* ASA I-III patients
* Age 18-50
* BMI ≤ 38 kg/m2

Exclusion Criteria:

* Refusal or inability to provide informed consent
* Any contraindication to regional anesthesia including coagulopathy or bleeding diathesis,
* Allergy to local anesthetics, or infection at the site of the block
* History of long-term opioid intake (more than 3 months use) or chronic pain disorder (more than 3 months)
* History of preexisting neuropathy in the operative leg
* Revision of ACL repair

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Oral morphine equivalent consumption | Up to 24-hours after surgery
  Cumulative oral morphine equivalent consumption over 24 hours post-op
Quadriceps motor strength | Pre-op, 30 minutes post-anesthesia
  Percent decrease in quadriceps motor strength at 30 minutes following anesthesia compared to baseline

SECONDARY OUTCOMES:
inta-operative opioid consumption | during surgery
  Cumulative amount of opioids consumed during surgery
Oral morphine equivalent consumption in PACU | PACU admission to PACU discharge (approximately 4 hours)
  Cumulative oral morphine equivalent consumed in PACU
Post-operative Pain | Up to 24 hours post-operative
  area under the curve for rest pain scores during the first 24 hours post-op, using the numeric pain rating scale from 0-10, with 0 being no pain and 10 being the worst possible pain
Quality of Recovery | At 24 hours post-operative
  Measured using the QoR-15 questionnaire at 24 hours post-op
Time in hospital | From hospital admission to hospital discharge (approximately 12 hours)
  Time from admission to discharge
Nerve Block Complications | up to 24 hours post-operative, up to 2 weeks post-operative
  Presence or absence of nerve block complications